CLINICAL TRIAL: NCT04317885
Title: A Study Evaluating Safety and Efficacy of C-CAR039 Treatment in Relapsed or Refractory NHL Subjects
Brief Title: A Study Evaluating Safety and Efficacy of C-CAR039 Treatment in NHL Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., Director, Department of Hematology, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-015
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-Hodgkin's B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prizloncabtagene Autoleucel (Experimental): Prizlon-cel will be intravenously administered as a single infusion after lymphodepletion
  Interventions: Biological: Prizloncabtagene Autoleucel

INTERVENTIONS:
Biological: Prizloncabtagene Autoleucel — Autologous 2nd generation CD19/CD20-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR039

SUMMARY:
The trial is a single arm, single-center, non-randomized phase I clinical trial which is designed to evaluate the safety and efficacy of C-CAR039 in treatment of relapsed or refractory NHL patients

DETAILED DESCRIPTION:
This study plans to enroll 25 patients to assess the safety and efficacy of C-CAR039. Subjects who meet the eligibility criteria will receive a single dose of C-CAR039 injection.

The study will include the following sequential phases: Screening, Apheresis and C-CAR039 manufacturing, Bridging (if needed), Baseline, lymphodepletion, C-CAR039 infusion, and Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteered to participate in this study and signed informed consent
* 2. Age 18-75 years old, male or female
* 3. CD19 or CD20 positive DLBCL (including PMBCL and tFL), FL and MCL confirmed by cytology or histology according to WHO2016 criteria. For CD20-positive subjects, they should have received at least one regimen containing anti-CD20-targeted therapy (such as rituximab). If they do not complete the regimen due to intolerance, the cause should be recorded.
* 4. Relapsed or refractory disease after ≥ 2 lines (for FL, at least 3 lines) of standard therapy or relapsed after autologous stem cell transplantation (ASCT)
* 5. At least one measurable lesion (LDi ≥ 1.5 cm);
* 6. At least two weeks from last treatment (radiation, chemotherapy, mAb, etc) to apheresis;
* 7. LVEF≥ 50% (ECHO)
* 8. No active pulmonary infections, normal or mild impaired pulmonary function and SpO2≥92%
* 9. Laboratory criteria: ANC≥1.0×109/L; Platelets≥50×109/L; Serum total bilirubin ≤1.5x ULN; Creatinine≤ ULN; AST and ALT≤3x ULN
* 10. No contraindications of apheresis;
* 11. Expected survival ≥ 3months
* 12. ECOG score 0 or 1

Exclusion Criteria:

* 1. Have a history of allergy to cellular products;
* 2. According to the NYHA cardiac function grading standards, patients with grade III or IV cardiac dysfunction;
* 3. A history of craniocerebral trauma, disturbance of consciousness, epilepsy, cerebrovascular ischemia, cerebrovascular hemorrhagic disease, etc.;
* 4. Patients with central nervous system involvement;
* 5. Patients with autoimmune diseases, immunodeficiency or other conditions requiring immunosuppressive therapy;
* 6. Received allogeneic hematopoietic stem cell transplantation before;
* 7. Previous use of any CAR T cell product or other genetically modified T cell therapy;
* 8. Autologous stem cell transplantation within 6 weeks before infusion;
* 9. Severe active infections (except for simple urinary tract infections, bacterial pharyngitis), or currently undergoing intravenous infusion of antibiotics. However, prophylactic antibiotic, antiviral and antifungal infection treatments are permissible;
* 10. Live vaccination within 4 weeks prior to apheresis;
* 11. People infected with HIV, HBV, HCV and TPPA/RPR, and carriers with HBV;
* 12. A history of alcohol abuse, drug use or mental illness;
* 13. Subjects who are not sterilized and have any of the following conditions:

  1. are pregnant/lactating; or
  2. planned pregnancy during the trial; or
  3. being fertile and unable to use effective contraception;
* 14. Severe hypersensitivity to fludarabine or cyclophosphamide;
* 15. A history of other primary cancers other than the following:

  1. Non-melanoma tumors such as basal cell carcinoma of the skin that are cured by excision
  2. Cured in situ cancers such as cervical, bladder, or breast cancer
* 16. The investigators consider that the subject has other conditions that are not suitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 12 weeks after C-CAR039 infusion
  Incidence and severity of adverse events after CAR-T infusion

SECONDARY OUTCOMES:
Overall Response rate (ORR) | Up to 24 Months after C-CAR039 infusion
  Complete response (CR) rate plus partial response (PR) rate by Lugano 2014 criteria
Duration of response (DOR) | Up to 24 Months after C-CAR039 infusion
  The time from the date of first response (PR or CR) to the date of disease progression or death after C-CAR039 infusion
Progression-free survival (PFS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of progression as assessed by Lugano 2014 criteria or death
Overall survival (OS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, MD, Ph.D, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu W, Li P, Zhou L, Yang M, Ye S, Zhu D, Huang J, Yao X, Zhang Y, Li L, Zhao J, Zhu K, Li J, Zheng C, Lan L, Wan H, Yao Y, Zhang H, Zhou D, Jin J, Liang A. A phase 1 trial of prizloncabtagene autoleucel, a CD19/CD20 CAR T-cell therapy for relapsed/refractory B-cell non-Hodgkin lymphoma. Blood. 2025 Apr 3;145(14):1526-1535. doi: 10.1182/blood.2024026401. PMID 39813680